CLINICAL TRIAL: NCT03254277
Title: A Phase 1 First-in-human Study of the Safety and Pharmacokinetics of 3BNC117-LS in HIV-infected and HIV-uninfected Individuals
Brief Title: 3BNC117-LS First-in-Human Phase 1 Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: YCO-0946
Record Dates: First submitted 2017-08-11; First posted 2017-08-18 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Human Immunodeficiency Virus
Keywords: Broadly Neutralizing Antibody; 3BNC117-LS; First in Human; Dose Escalation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Antibodies, Monoclonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Group 1A (Experimental): HIV-uninfected individuals will be administered one infusion of 3BNC117-LS dosed at 3 mg/kg.
  Interventions: Drug: 3BNC117-LS
- Group 1B (Experimental): HIV-uninfected individuals will be administered one infusion of 3BNC117-LS dosed at 10 mg/kg.
  Interventions: Drug: 3BNC117-LS
- Group 1C (Experimental): HIV-uninfected individuals will be administered one infusion of 3BNC117-LS dosed at 30 mg/kg.
  Interventions: Drug: 3BNC117-LS
- Group 2B (Experimental): HIV-infected individuals on ART with HIV-1 plasma RNA levels < 20 copies/ml or off ART for at least 8 weeks with HIV-1 plasma RNA levels < 100,000 copies/ml, will be administered one infusion of 3BNC117-LS dosed at 10 mg/kg.
  Interventions: Drug: 3BNC117-LS
- Group 2C (Experimental): HIV-infected individuals on ART with HIV-1 plasma RNA levels < 20 copies/ml, or off ART for at least 8 weeks with HIV-1 plasma RNA levels < 100,000 copies/ml, will be administered one infusion of 3BNC117-LS dosed at 30 mg/kg.
  Interventions: Drug: 3BNC117-LS
- Group 1D (Experimental): HIV-uninfected individuals will be administered one infusion of 3BNC117-LS dosed at 30 mg/kg.
  Interventions: Drug: 3BNC117-LS
- Group 2D (Experimental): HIV-infected individuals on ART with HIV-1 plasma RNA levels < 20 copies/ml will be administered one infusion of 3BNC117-LS dosed at 30 mg/kg.
  Interventions: Drug: 3BNC117-LS
- Group 1E (Experimental): HIV-uninfected individuals will be administered a single 1 mL (approximately 150 mg) subcutaneous injection of 3BNC117-LS or placebo in a 3:1 ratio.
  Interventions: Drug: 3BNC117-LS; Drug: Placebo
- Group 1F (Experimental): HIV-uninfected individuals will be administered a single 2 mL (approximately 300 mg) subcutaneous injection of 3BNC117-LS or placebo in a 3:1 ratio.
  Interventions: Drug: 3BNC117-LS; Drug: Placebo

INTERVENTIONS:
Drug: 3BNC117-LS — Intravenous infusion of 3BNC117-LS
  Other Names: Monoclonal Antibody
Drug: Placebo — Placebo
  Arms: Group 1E; Group 1F

SUMMARY:
The proposed study is a phase 1 study of the mAb 3BNC117-LS administered intravenously in HIV uninfected individuals and HIV-infected individuals, and subcutaneously in HIV-uninfected individuals.The objectives of the study are to evaluate the safety, tolerability and pharmacokinetics of a single administration of 3BNC117-LS.

DETAILED DESCRIPTION:
The proposed study is a Phase 1, open label, dose escalation cohort study of 3BNC117-LS administered intravenously in HIV-uninfected and HIV-1 infected participants.

This study consists of two parts. In part A, study participants will be enrolled in an open label manner to receive a single intravenous infusion of 3BNC117-LS at one of three increasing dose levels (3 mg/kg, 10 mg/kg and 30 mg/kg). Participants in Part B will also receive a single administration of 3BNC117-LS, however, the product administered in Part B of the study derives from a new manufacturing lot. The manufacturing lot used in Part A had incomplete glycosylation of the 3BNC117-LS light chain, which has been corrected in the new lot. Participants in Part B will receive 3BNC117-LS intravenously at 30 mg/kg in an open label manner (HIV-uninfected and HIV-infected) or will be randomized to receive a subcutaneous injection of 3BNC117-LS or placebo in a double-blinded fashion (HIV-uninfected only).

Part A has already been enrolled with 21 participants. Part B has a planned enrollment of 22 participants.

Part A

* Group 1A (n=3-6) - HIV-uninfected individuals will be administered one infusion of 3BNC117-LS dosed at 3 mg/kg.
* Group 1B (n=3-6) - HIV-uninfected individuals will be administered one infusion of 3BNC117-LS dosed at 10 mg/kg.
* Group 1C (n=3-6) - HIV-uninfected individuals will be administered one infusion of 3BNC117-LS dosed at 30 mg/kg.
* Group 2B (n=6) - HIV-infected individuals on ART with HIV-1 plasma RNA levels < 20 copies/ml or off ART for at least 8 weeks with HIV-1 plasma RNA levels < 100,000 copies/ml, will be administered one infusion of 3BNC117-LS dosed at 10 mg/kg.
* Group 2C (n=6) - HIV-infected individuals on ART with HIV-1 plasma RNA levels < 20 copies/ml, or off ART for at least 8 weeks with HIV-1 plasma RNA levels < 100,000 copies/ml, will be administered one infusion of 3BNC117-LS dosed at 30 mg/kg.

Part B

* Group 1D (n=3) - HIV-uninfected individuals will be administered one infusion of 3BNC117-LS dosed at 30 mg/kg.
* Group 2D (n=3) - HIV-infected individuals on ART with HIV-1 plasma RNA levels < 20 copies/ml will be administered one infusion of 3BNC117-LS dosed at 30 mg/kg.
* Group 1E (n=8) - HIV-uninfected individuals will be administered a single 1 mL (approximately 150 mg) subcutaneous injection of 3BNC117-LS or placebo in a 3:1 ratio.
* Group 1F (n=8) - HIV-uninfected individuals will be administered a single 2 mL (approximately 300 mg) subcutaneous injection of 3BNC117-LS or placebo in a 3:1 ratio.

Following 3BNC117-LS infusion, study participants will return for safety assessments at weeks 1, 2 and 4 following infusion, then bi-monthly or monthly until the end of study follow up.

Serum samples for PK (pharmacokinetic) measurements will be collected before 3BNC117-LS infusion, at the end of the infusion, and at multiple time points during study follow up.

Samples will also be collected for measurement of HIV-1 plasma RNA levels before 3BNC117-LS infusion (screen, pre-infusion and day 0) and at all follow up visits in Groups 2B and 2C.

All participants will be followed for 48 weeks after 3BNC117-LS administration.

ELIGIBILITY:
Inclusion Criteria:

Groups 1A-1F (HIV-uninfected):

1. Males and females, age 18 to 65
2. Amenable to HIV risk reduction counseling and agrees to maintain behavior consistent with low risk of HIV exposure.
3. If sexually active male or female, and participating in sexual activity that could lead to pregnancy, agrees to use two effective methods of contraception (i.e. condom with spermicide, diaphragm with spermicide, hormone-eluting IUD, hormone-based contraceptive with condom) from 10 days prior to and until seven months after 3BNC117-LS infusion, and agrees to safer sex counseling at each visit.

   * Female study participants of reproductive potential are defined as pre-menopausal women who have not had a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, tubal ligation or salpingectomy). Women are considered menopausal if they have not had a menses for at least 12 months and have a FSH of greater than 40 IU/L or if FSH testing is not available, they have had amenorrhea for 24 consecutive months.

Groups 2B-2D (HIV-infected):

1. Males and females, age 18 to 65.
2. HIV-1 infection confirmed by two laboratory assays.
3. HIV-infected individuals off ART for at least 8 weeks with HIV-1 plasma RNA levels < 100,000 copies/ml by standard assays (ART-naïve or off ART due to intolerance or by choice), or on ART with HIV-1 plasma RNA levels < 20 copies/ml. HIV-1 RNA levels should be measured on 2 occasions, at least 1 week apart. At least one measurement must be performed within 49 days prior to enrollment (day 0). Group 2D will only enroll HIV-infected individuals on ART.
4. Current CD4+ T cell count > 300 cells/μl.
5. If sexually active male or female, and participating in sexual activity that could lead to pregnancy or transmission of HIV, agrees to use two effective methods of contraception (i.e. condom with spermicide, diaphragm with spermicide, hormone-eluting IUD, hormone-based contraceptive with condom) from 10 days prior to and until seven months after 3BNC117-LS infusion, and agrees to safer sex counseling at each visit.

Exclusion Criteria:

Groups 1A-1F (HIV-uninfected):

1. Confirmed HIV-1 or HIV-2 infection.
2. History of immunodeficiency or autoimmune disease; use of systemic corticosteroids, immunosuppressive anti-cancer, or other medications considered significant by the trial physician within the last 6 months.
3. Any clinically significant acute or chronic medical condition (such as autoimmune diseases) that in the opinion of the investigator would preclude participation.
4. Within the 12 months prior to enrollment, the participant has a history of sexually transmitted infection.
5. Hepatitis B or C infection as indicated by the presence of Hepatitis B surface antigen (HBsAg) or hepatitis C virus RNA (HCV-RNA) in blood.
6. Laboratory abnormalities in the parameters listed:

   * Absolute neutrophil count ≤ 1,500 cells/µL;
   * Hemoglobin ≤ 11 gm/dL if female; ≤ 12.5 gm/dL if male;
   * Platelet count ≤ 125,000 cells/µL;
   * Alanine transaminase (ALT) ≥ 1.25 x ULN;
   * Aspartate transaminase (AST) ≥ 1.25 x ULN;
   * Alkaline phosphatase ≥ 1.5 x ULN;
   * Total bilirubin > 1 x ULN;
   * Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73m2.
7. Pregnancy or lactation.
8. Any vaccination within 14 days prior to 3BNC117-LS infusion.
9. Receipt of any experimental HIV vaccine or monoclonal antibody therapy of any kind in the past.
10. History of severe reaction to a vaccine or drug infusion or history of severe allergic reactions.
11. Individuals with known hypersensitivity to any constituent of the investigational product.
12. Receipt of another investigational product currently or within the past 12 weeks, or expected concurrent participation in another study in which investigational products will be administered.

Groups 2B-2D (HIV-infected):

1. Have a history of AIDS-defining illness within 3 years prior to enrollment.
2. History of systemic corticosteroids, immunosuppressive anti-cancer, or other medications considered significant by the trial physician within the last 6 months.
3. Any clinically significant acute or chronic medical condition (such as autoimmune diseases), other than HIV infection, that in the opinion of the investigator would preclude participation.
4. Hepatitis B or C infection as indicated by the presence of Hepatitis B surface antigen (HBsAg) or hepatitis C virus RNA (HCV-RNA) in blood.
5. Laboratory abnormalities in the parameters listed below:

   * Absolute neutrophil count ≤ 1,000 cells/μl;
   * Hemoglobin ≤ 10 gm/dL;
   * Platelet count ≤ 100,000 cells/μl;
   * ALT ≥ 1.5 x ULN;
   * AST ≥ 1.5 x ULN;
   * Alkaline phosphatase ≥ 1.5 x ULN;
   * Total bilirubin > 1 x ULN;
   * eGFR < 60 mL/min/1.73m2.
6. Pregnancy or lactation.
7. Any vaccination within 14 days prior to 3BNC117-LS infusion.
8. Receipt of any experimental HIV vaccine or monoclonal antibody therapy of any kind in the past.
9. History of severe reaction to a vaccine or drug infusion or history of severe allergic reactions.
10. Individuals with known hypersensitivity to any constituent of the investigational product.
11. Receipt of another investigational product currently or within the past 12 weeks, or expected concurrent participation in another study in which investigational products will be administered.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
The number of participants who experience adverse events within 2 weeks after 3BNC117-LS infusion in all study groups | 2 weeks following the 3BNC117-LS infusion
  Adverse events include signs, symptoms and laboratory abnormalities, in addition to local and systemic reactogenicity adverse events.
Elimination half-life (t1/2) of 3BNC117-LS in all study groups | 48 weeks
  Elimination half-life (t1/2) of 3BNC117-LS in all study groups
Clearance (CL/F) of 3BNC117-LS in all study groups | 48 weeks
  Clearance (CL/F) of 3BNC117-LS in all study groups
Volume of distribution (Vz/F) of 3BNC117-LS in all study groups | 48 weeks
  Volume of distribution (Vz/F) of 3BNC117-LS in all study groups
Area under the curve of 3BNC117-LS in all study groups | 48 weeks
  Area under the curve of 3BNC117-LS in all study groups
Decay curve of 3BNC117-LS in all study groups | 48 weeks
  Decay curve of 3BNC117-LS in all study groups

SECONDARY OUTCOMES:
Frequency of induced anti-3BNC117-LS antibodies in all study groups. | 48 weeks
  Frequency of induced anti-3BNC117-LS antibodies in all study groups.
Levels of induced anti-3BNC117-LS antibodies in all study groups. | 48 weeks
  Levels of induced anti-3BNC117-LS antibodies in all study groups.
The number of participants who experience adverse events during study follow-up | 48 weeks
  Adverse events include signs, symptoms and laboratory abnormalities

OTHER OUTCOMES:
3BNC117-LS levels in cervicovaginal and rectal fluids | Day 0 and 2 weeks following 3BNC117-LS infusion
  3BNC117-LS levels in cervicovaginal and rectal fluids
The decline in plasma HIV-1 RNA level after 3BNC117-LS infusion in viremic HIV-infected individuals | 48 weeks
  The decline in plasma HIV-1 RNA level after 3BNC117-LS infusion in viremic HIV-infected individuals
Analysis of escape viruses in individuals not on ART | 48 weeks
  Phenotypic and genotypic analysis of escape viruses in individuals not on ART.
Levels of cell-associated HIV-1 RNA and DNA before and after 3BNC117-LS infusion. | 48 weeks
  Levels of cell-associated HIV-1 RNA and DNA before and after 3BNC117-LS infusion.
Serum neutralizing activity against a panel of HIV-1 isolates before and after 3BNC117-LS infusion. | 48 weeks
  Serum neutralizing activity against a panel of HIV-1 isolates before and after 3BNC117-LS infusion.
HIV-specific T and B cell immune responses following 3BNC117-LS infusion | 48 weeks
  HIV-specific T and B cell immune responses following 3BNC117-LS infusion
T cell counts after 3BNC117-LS infusion | 48 weeks
  Absolute and relative CD4 + and CD8+ T cell counts after 3BNC117-LS infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Caskey, MD, Principal Investigator — The Rockefeller University
Locations (1):
- The Rockefeller University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Valente PK, Wu Y, Cohen YZ, Caskey M, Meyers K. Behavioral and social science research to support development of educational materials for clinical trials of broadly neutralizing antibodies for HIV treatment and prevention. Clin Trials. 2021 Feb;18(1):17-27. doi: 10.1177/1740774520948042. Epub 2020 Aug 24. PMID 32838558